CLINICAL TRIAL: NCT02268669
Title: A Randomized Clinical Trial Comparing Primary PCI and Post-thrombolysis PCI as Reperfusion Strategies in Patients With ST Segment Elevation Acute Myocardial Infarction
Brief Title: Comparison of Primary PCI vs. Post-thrombolysis PCI as Reperfusion Strategies in STEMI
Acronym: GRACIA4
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GRACIA Group (Other)
Responsible Party: Principal Investigator, Pedro L Sanchez, Coordinator, GRACIA Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRACIA4
Record Dates: First submitted 2014-10-13; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Myocardial Infarction
Keywords: primary angioplasty; post-thrombolysis angioplasty; ST elevation acute myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary angioplasty (Active Comparator): Patients assigned to this treatment will undergo cardiac catheterization within the time recommended by current guidelines. Double antiagregation will be used, vascular access wil be obtained and bivalirudin will be used as anticoagulation; all following current guidelines recommendations
  Interventions: Other: Reperfusion strategies
- Post-thrombolysis angioplasty (Active Comparator): Patients will receive tenecteplase, enoxaparin, and double antiagreagation with clopidogrel or aspirin as recommended guidelines. Criteria of no reperfusion after fibrinolysis is defined as absence of ST-segment lowering >50%, 90 minutes after fibrinolysis. If not reperfusion is achieved recue angiplasty will be performed inmmediately if reperfusion is achieved cardiac catheterization will be performed the mornig following the day of randomization
  Interventions: Other: Reperfusion strategies

INTERVENTIONS:
Other: Reperfusion strategies — Two different reperfusion strategies in STEMI will be compared: primary angioplasty vs. post-thrombolysis angioplasty

SUMMARY:
The conceptual hypothesis of this study is that primary angioplasty is superior to a combined strategy of immediate thrombolysis followed by routine angioplasty in patients with ST-segment elevation acute myocardial infarction (STEMI), even with the inherent delay of the transfer of these patients.

DETAILED DESCRIPTION:
This is a randomized, multicenter, open-label clinical trial comparing two strategies of reperfusion in STEMI. Patients will be randomly allocated to: primary angioplasty or post-thrombolysis angioplasty. A clinical follow-up will be performed at 12 months. In this trial, 1444 patients with STEMI will be randomized to primary angioplasty with immediate stent implantation in at least the infarct related artery (IRA) under bivalirudin protection, or to a combined strategy of immediate thrombolysis with tenecteplase (TNK) and enoxaparin followed by cardiac catheterization and adequate revascularization when indicated during the next morning after randomization.

Primary endpoint:

To compare the clinical efficacy (incidence of the composite endpoint formed by death, reinfarction, new revascularization, rehospitalization or severe hemorrhage within 12 months) of primary angioplasty versus thrombolytic treatment followed by percutaneous coronary intervention (PCI) the next day in patients with STEMI.

Secondary endpoints:

* Components of the composite endpoint individually analysed at 12 months (death, reinfarction, new revascularization, rehospitalization and severe hemorrhage).
* Cardiovascular mortality and its different components (pre-specified in the case report forms, CRF) at 12 months.
* Incidence of the composite endpoint formed by death, reinfarction, new revascularization, rehospitalization and/or hemorrhage at 30 days.
* Incidence of major bleeding events during hospitalization and at 30 days.
* To compare the clinical efficacy of both treatments according to the timing of presentation after symptom onset (0 to 3 hours, >3-6 hours, and >6-12 hours), to the patient´s age (> or < 75 years), to the infarction localization (anterior or inferior), to gender (male or female), to the presence of diabetes mellitus and to the characteristics of the recruiting center (with or without 24-hour catheterization facilities).
* Incidence of the composite endpoint formed by death, reinfarction, new revascularization, rehospitalization and/or hemorrhage at 3 years.
* Components of the composite endpoint individually analysed at 3 years (death, reinfarction, new revascularization, rehospitalization and severe hemorrhage).
* Analysis of stent thrombosis according to the Academic Research Consortium (ARC) definition (http://www.fda.gov/ohrms/dockets/ac/06/transcripts/2006-4253t2.rtf.) within 30 days, 12 months and 3 years.
* To compare the combination of death, reinfarction, revascularization, rehospitalization and/or major hemorrhage of patients treated with primary angioplasty versus those assigned to the postrombolysis angioplasty who underwent catheterization the following day within 30 days, 12 months and 3 years.
* To compare every indivicual components of the combine endpoint (death, reinfarction, revascularization, rehospitalization and major hemorrhage) of patients treated with primary angioplasty versus those assigned to the postrombolysis angioplasty who underwent catheterization the following day within 30 days, 12 months and 3 years.
* To compare the cost-effectiveness relationship (cost of maintaining a patient alive and without adverse cardiovascular events within the first year post-infarction) of both strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Chest discomfort > 30 minutes with no response to nitroglycerin
* Time from the onset of symptoms to randomization between 0 and 12 hours
* ST segment elevation > 1 mm in two or more contiguos precordial leads or non-diagnostic ECG (left bundle branch block or pacemarker rhythm) with classic symptoms.
* Killip class equal or less than 3
* Written informed consent

Exclusion Criteria:

* Cardiogenic shock defined as a systolic blood pressure <90 mm Hg without response to fluid administration or <100 mm Hg in patients with supportive treatment and no bradycardia
* Suspicion or evidence of mechanical complications of STEMI
* Non-cardiac disease that is likely to jeopardize compliance with follow-up schedule of the study (life expectancy < 1 year)
* woman of childbearing potential unless a negative pregnant test
* Major contraindications for thrombolytic therapy
* Participation in other trial
* Known multivessel disease identified as unsuitable for revascularization
* Known peripheral vascular disease that complicates cardiac catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1444 (Actual)
Dates: Start 2010-05; Primary Completion 2014-10 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
incidence of the composite endpoint formed by death, reinfarction, new revascularization, rehospitalization or severe hemorrhage | 12 months
  To compare the clinical efficacy (incidence of the composite endpoint formed by death, reinfarction, new revascularization, rehospitalization or severe hemorrhage within 12 months) of primary angioplasty versus post-thrombolytic angioplasty

SECONDARY OUTCOMES:
Incidence of death | 12 months
  Components of the composite endpoint individually analysed at 12 months (death, reinfarction, new revascularization, rehospitalization and severe hemorrhage).
Incidence of myocardial reinfaction | 12 months
  Components of the composite endpoint individually analysed at 12 months (death, reinfarction, new revascularization, rehospitalization and severe hemorrhage).
Incidence of new revascularization | 12 months
  Components of the composite endpoint individually analysed at 12 months (death, reinfarction, new revascularization, rehospitalization and severe hemorrhage).
Incidence of rehospitalization | 12 months
  Components of the composite endpoint individually analysed at 12 months (death, reinfarction, new revascularization, rehospitalization and severe hemorrhage).
Incidence of cardiovascular mortality | 12 months
Incidence of the composite endpoint formed by death, reinfarction, new revascularization, rehospitalization and/or hemorrhage | 30 days
Incidence of major bleeding events | Hospitalization and at 30 days
clinical efficacy according to timing of presentation (<3, 3-6, and >6 hours), patient´s age (> or < 75 years), infarction localization, gender, presence of diabetes and recruiting center (with or without catheterization facilities) | 12 months
Incidence of the composite endpoint formed by death, reinfarction, new revascularization, rehospitalization and/or hemorrhage | 3 years
Incidence of death | 3 years
Incidence of reinfarction | 3 years
Incidence of new revascularization | 3 years
Incidence of rehospitalization | 3 years
Analysis of stent thrombosis according to the Academic Research Consortium (ARC) definition (http://www.fda.gov/ohrms/dockets/ac/06/transcripts/2006-4253t2.rtf.) | 30 days, 12 months and 3 years
Combination of death, reinfarction, revascularization, rehospitalization and/or major hemorrhage of patients treated with primary angioplasty vs. those assigned to postrombolysis angioplasty undergoing catheterization the following day | 30 days, 12 months and 3 years
To compare every indivicual components of the combine endpoint of patients treated with primary angioplasty versus those assigned to the postrombolysis angioplasty who underwent catheterization the following day | 30 days, 12 months and 3 years
To compare the cost-effectiveness relationship (cost of maintaining a patient alive and without adverse cardiovascular events within the first year post-infarction) of both strategies | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Fernandez-Aviles, MD, PhD, Study Chair — faviles@secardiologia.es

REFERENCES:
- [Background] Fernandez-Aviles F, Alonso JJ, Castro-Beiras A, Vazquez N, Blanco J, Alonso-Briales J, Lopez-Mesa J, Fernandez-Vazquez F, Calvo I, Martinez-Elbal L, San Roman JA, Ramos B; GRACIA (Grupo de Analisis de la Cardiopatia Isquemica Aguda) Group. Routine invasive strategy within 24 hours of thrombolysis versus ischaemia-guided conservative approach for acute myocardial infarction with ST-segment elevation (GRACIA-1): a randomised controlled trial. Lancet. 2004 Sep 18-24;364(9439):1045-53. doi: 10.1016/S0140-6736(04)17059-1. PMID 15380963
- [Background] Fernandez-Aviles F, Alonso JJ, Pena G, Blanco J, Alonso-Briales J, Lopez-Mesa J, Fernandez-Vazquez F, Moreu J, Hernandez RA, Castro-Beiras A, Gabriel R, Gibson CM, Sanchez PL; GRACIA-2 (Groupo de Analisis de Cardiopatia Isquemica Aguda) Investigators. Primary angioplasty vs. early routine post-fibrinolysis angioplasty for acute myocardial infarction with ST-segment elevation: the GRACIA-2 non-inferiority, randomized, controlled trial. Eur Heart J. 2007 Apr;28(8):949-60. doi: 10.1093/eurheartj/ehl461. Epub 2007 Jan 23. PMID 17244641
- [Background] Sanchez PL, Gimeno F, Ancillo P, Sanz JJ, Alonso-Briales JH, Bosa F, Santos I, Sanchis J, Bethencourt A, Lopez-Messa J, de Prado AP, Alonso JJ, San Roman JA, Fernandez-Aviles F. Role of the paclitaxel-eluting stent and tirofiban in patients with ST-elevation myocardial infarction undergoing postfibrinolysis angioplasty: the GRACIA-3 randomized clinical trial. Circ Cardiovasc Interv. 2010 Aug;3(4):297-307. doi: 10.1161/CIRCINTERVENTIONS.109.920868. PMID 20716757